CLINICAL TRIAL: NCT06140771
Title: A Three-Month Clinical Study to Assess the Gingivitis Effects of Various Dentifrices
Brief Title: A Clinical Study to Assess the Gingivitis Effects of Various Dentifrices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021080
Record Dates: First submitted 2023-11-14; First posted 2023-11-20 (Actual); Last update posted 2023-11-20 (Actual); Status verified 2023-11

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.76% Sodium Monofluorophosphate Dentifrice (Sham Comparator)
  Interventions: Drug: 0.76% Sodium Monofluorophosphate Dentifrice
- 1.15% Sodium Monofluorophosphate Dentifrice (Sham Comparator)
  Interventions: Drug: 1.15% Sodium Monofluorophosphate Dentifrice
- Marketed 0.454% Stannous Fluoride Dentifrice (Active Comparator)
  Interventions: Drug: 0.454% Stannous Fluoride Dentifrice
- 0.454% Stannous Fluoride Dentifrice (Active Comparator)
  Interventions: Drug: 0.454% Stannous Fluoride Dentifrice

INTERVENTIONS:
Drug: 0.76% Sodium Monofluorophosphate Dentifrice — Whole mouth brushing with a toothpaste, twice daily for the duration of the study.
  Arms: 0.76% Sodium Monofluorophosphate Dentifrice
Drug: 1.15% Sodium Monofluorophosphate Dentifrice — Whole mouth brushing with a toothpaste, twice daily for the duration of the study.
  Arms: 1.15% Sodium Monofluorophosphate Dentifrice
Drug: 0.454% Stannous Fluoride Dentifrice — Whole mouth brushing with a toothpaste, twice daily for the duration of the study.
  Arms: Marketed 0.454% Stannous Fluoride Dentifrice
Drug: 0.454% Stannous Fluoride Dentifrice — Whole mouth brushing with a toothpaste, twice daily for the duration of the study.
  Arms: 0.454% Stannous Fluoride Dentifrice

SUMMARY:
The objective of this learning clinical study is to assess the gingivitis effects of four different dentifrices over a 3-month period.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* Be in general good health as determined by the Investigator based on a review of the health history/update for participation in the trial;
* Have at least 16 gradable teeth;
* Have mild to moderate gingivitis with a range of 10% to 70% bleeding sites;
* Agree to return for scheduled visits and follow the study procedures;
* Agree to refrain from use of any non-study oral hygiene products for the duration of the study;
* Agree to delay any elective dentistry, including dental prophylaxis, until the completion of the study.

Exclusion Criteria:

* Having taken antibiotic, anti-inflammatory, or anti-coagulant medications within 4 weeks of the Baseline Visit;
* Have any oral conditions that could interfere with study compliance and/or examination procedures, such as widespread caries, soft or hard tissue tumor of the oral cavity, or advanced periodontal disease;
* Removable oral appliances;
* Fixed facial or lingual orthodontic appliances;
* Self-reported pregnancy or lactation;
* Any diseases or condition that might interfere with the safe participation in the study; and
* Inability to undergo study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-02-06 (Actual); Study Completion 2022-02-06 (Actual)

PRIMARY OUTCOMES:
Löe-Silness Gingivitis Evaluation | 3 Months
  Löe-Silness Gingivitis Evaluation is a validated assessment of gingival health looking at inflammation and bleeding based on a 4 point range 0 (normal gingiva) to 3 (severe inflammation).

SECONDARY OUTCOMES:
Löe-Silness Gingivitis Evaluation | Baseline
  Löe-Silness Gingivitis Evaluation is a validated assessment of gingival health looking at inflammation and bleeding based on a 4 point range 0 (normal gingiva) to 3 (severe inflammation).
Löe-Silness Gingivitis Evaluation | 1 Month
  Löe-Silness Gingivitis Evaluation is a validated assessment of gingival health looking at inflammation and bleeding based on a 4 point range 0 (normal gingiva) to 3 (severe inflammation).

CONTACTS AND LOCATIONS:
Locations (1):
- UHRG, Whittier, California, United States